CLINICAL TRIAL: NCT00649870
Title: Single-Dose Food In Vivo Bioequivalence Study of Valacyclovir Hydrochloride Tablets (1000 mg; Mylan) to Valtrex® Tablets (1000 mg; GlaxoSmithKline) in Healthy Volunteers
Brief Title: Food Study of Valacyclovir Hydrochloride Tablets 1000 mg to Valtrex® Tablets 1000 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Wayne Talton, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: VALA-0405
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Valacyclovir

ARMS (2):
- 1 (Experimental): Valacyclovir Hydrochloride Tablets 1000 mg
  Interventions: Drug: Valacyclovir Hydrochloride Tablets 1000 mg
- 2 (Active Comparator): Valtrex® Tablets 1000 mg
  Interventions: Drug: Valtrex® Tablets 1000 mg

INTERVENTIONS:
Drug: Valacyclovir Hydrochloride Tablets 1000 mg — 1000mg, single dose fed
  Arms: 1
Drug: Valtrex® Tablets 1000 mg — 1000mg, single dose fed
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's valacyclovir hydrochloride 1000 mg tablets to GlaxoSmithKline's Valtrex® 1000 mg tablets following a single, oral 1000 mg (1 x 1000 mg) dose administration under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy, adult subjects, 18 years and older
* able to swallow medication

Exclusion Criteria:

* institutionalized subjects
* history of any significant disease
* use of any prescription or OTC medications within 14 days of start of study
* received any investigational products within 30 days prior to start of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-05; Primary Completion 2005-05 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
The 90% confidence interval for the LSMeans ratio of CPEAK, AUCL, and AUCI for the test and reference product should be between 80.00% and 125.00% for the natural log-transformed data. | blood collections through 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Williams, M.D., Principal Investigator — Kendle International Inc.
Locations (1):
- Kendle International Inc., Morgantown, West Virginia, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html